CLINICAL TRIAL: NCT07155876
Title: Exploring the Effect of Aromatherapy Inhalation for Managing Pain, Anxiety, and Nausea/Vomiting Throughout the Laboring Process
Brief Title: Exploring the Effect of Aromatherapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2298893
Record Dates: First submitted 2025-08-14; First posted 2025-09-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Labor Pain; Nausea and Vomiting
MeSH Terms: conditions — Anxiety Disorders; Labor Pain; Nausea; Vomiting | interventions — Aromatherapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Education video (Experimental): The participant receives aromatherapy plus standard of care (SoC) for treatment based on symptoms (anxiety, pain, and/or nausea/vomiting) as prescribed by the physician.
  Interventions: Other: Aromatherapy plus standard of care
- Control group: Standard of Care (Other): The patient receives SoC for treatment of based on symptoms (anxiety, pain, and/or nausea/vomiting) as prescribed by the physician.
  Interventions: Other: Standard of Care Only

INTERVENTIONS:
Other: Aromatherapy plus standard of care — The participant is offered an aromatherapy scented tab that is attached to their gown based on symptoms (anxiety, pain, and/or nausea/vomiting):
  1. Pain or anxiety: lavender or lavender sandalwood,
  2. Nausea/vomiting: orange ginger, or
  3. Despite the type of discomfort, the participant may request the alternate scent if the scent offered is not to their liking.
  Plus, the patient receives SoC for treatment based on symptoms (anxiety, pain, and/or nausea/vomiting) as prescribed by the physician.
  Arms: Intervention group: Education video
Other: Standard of Care Only — Participant receives symptom management medications for pain, nausea/vomiting, and/or anxiety as prescribed by the physician.
  Arms: Control group: Standard of Care

SUMMARY:
To explore the effect of aromatherapy in laboring patients with pain, anxiety, and/or nausea/vomiting.

ELIGIBILITY:
Inclusion Criteria:

• Pregnant patients at least 18 years old in spontaneous labor or induction of labor (despite transitioning into a caesarean section)

Exclusion Criteria:

* Patients who are unable to detect scents/odors
* Patients with known allergies to aromatherapy and/or its components

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Relief of nausea/vomiting | Measured before and after receiving standard of care (SoC) or Intervention+SoC.
  Measured in the control and intervention groups before and after receiving treatment (yes or no - presence of nausea/vomiting).
Decreased anxiety | Measured before and after receiving standard of care (SoC) or Intervention+SoC.
  Measured before and after receiving treatment in both the control and intervention groups. Anxiety level = 0 =none, 1 = minimal (a little), 2 = moderate (medium), and 3 = severe (a lot).
Pain relief (scale of 0 to 10) | Measured before and after receiving standard of care (SoC) or Intervention+SoC.
  Level of pain is measured before and after receiving treatment in both the control and interventions groups. Pain is measured on a scale of 0 to 10 (0 = no pain, 10 = severe pain).

CONTACTS AND LOCATIONS:
Locations (1):
- South Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No